CLINICAL TRIAL: NCT02262611
Title: Post Marketing Surveillance Study in Rehabilitation Clinics (Cardio, Nephro, Diabetes, Pulmo)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.428; 502.429, 502.430, 502.431 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; telmisartan, hydrochlorothiazide drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Hypertension patients - Pneumology
  Interventions: Drug: Micardis®; Drug: MicardisPlus®
- Hypertension patients - Cardiology
  Interventions: Drug: Micardis®; Drug: MicardisPlus®
- Hypertension patients - Nephrology
  Interventions: Drug: Micardis®; Drug: MicardisPlus®
- Hypertension patients - Diabetology
  Interventions: Drug: Micardis®; Drug: MicardisPlus®

INTERVENTIONS:
Drug: Micardis®
Drug: MicardisPlus®

SUMMARY:
Study to obtain long-term data on effects, safety and tolerability in routine medical practice and to investigate the potential of telmisartan to prevent secondary organ damage

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both gender aged >=18 admitted to a hospital due to insufficiently controlled essential hypertension.

No additional selection criteria have to be considered. Treatment was at the discretion of the physician following the summary of product information for Micardis® and MicardisPlus®

Exclusion Criteria:

* not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension recruited at hospitals in Germany specialized in cardiology, nephrology, diabetology and pneumology
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 1 year
Number of patients with abnormal changes in laboratory parameters | up to 1 year
Number of patients with clinically significant changes in vital signs | up to 1 year
Change in systolic blood pressure | up to 1 year
Change in diastolic blood pressure | up to 1 year

SECONDARY OUTCOMES:
Global assessment of efficacy by investigator on a 4-point scale | 2 weeks, after 1 year
Global assessment of tolerability by investigator on a 4-point scale | 2 weeks, after 1 year